CLINICAL TRIAL: NCT05044858
Title: Analgesic Efficacy of Pre-emptive Ultrasound-Guided Mid-Point Transverse Process to Pleura Block for Patients Undergoing Posterolateral Thoracotomy Incisions: Randomized Controlled Trial
Brief Title: Ultrasound-Guided Mid-Point Transverse Process to Pleura Block for Thoracotomy Incisions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Abdelhamid Mohamed, Resident of Anesthesiology and Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34646/4/21
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Pre-emptive; Postoperative Pain; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midpoint transverse process block group (Experimental): Patients will receive midpoint transverse process block after induction of general anesthesia and before surgical incision
  Interventions: Procedure: Midpoint transverse process block group
- Sham group (Sham Comparator): Patients will receive general anesthesia and the same intervention steps will be performed i.e., the block under investigation but instead of local anesthetic a placebo (2ml normal saline) will be injected (sham block)
  Interventions: Procedure: Sham group

INTERVENTIONS:
Procedure: Midpoint transverse process block group — After marking the level of the incision by surgeon (commonly T5- T6) The patient will be situated in the lateral position, the block area will be sterilized with povidine-iodine, and high -frequency linear ultrasound probe will be placed oblique parasagittally 3 cm lateral to the spinous process at the level of skin incision. 100-mm short bevel echogenic needle (Contiplex, B.Braun, Germany) will be inserted in plane from cranial to caudal direction. The desired end point of the needle tip will be the midpoint of the line between the posterior border of transverse process and the pleura titrated bolus of 20 ml of 0.25% bupivacaine and dexamethazone 8 mg will be injected at the target site. At end of the surgery general anaesthesia will be stopped with reversal of muscle relaxation and awakening of patient
  Arms: Midpoint transverse process block group
Procedure: Sham group — General anesthesia will be induced with the same protocol and MTP block will be done but with injection of placebo (2 ml normal saline) instead of local anesthetic .
  On arrival to the PACU postoperative Numerical Rating scale at rest and coughing will be recorded, analgesia will be maintained with intravenous paracetamol 1 g every 8 h and required additional rescue analgesia (morphine) at any time will be calculated.
  Arms: Sham group

SUMMARY:
This study is designed to investigate the analgesic efficacy of pre-emptive ultrasound-guided midpoint transverse process to pleura (MTP) block for posterolateral thoracotomy in cardiothoracic surgeries.

DETAILED DESCRIPTION:
Preemptive preoperative analgesia was first proposed, over the years it has been gradually regarded as an intervention given before incision, facilitating mobilization and functional rehabilitation after surgery, reducing postoperative opioid consumption, decreasing the incidence of adverse events and improving patient satisfaction.

The Mid Transverse Process to Pleura block, described by Costach et al. involves deposition of drug midway between the transverse process and pleura. Costach et al. postulated that the local anesthetic deposited at this point may reach the paravertebral space through several possible mechanisms, such as spread medially through the gap between the superior costotransverse ligament (SCTL) and vertebral bodies, through fenestrations in SCTL, and laterally through the internal intercostal membrane

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21- and65 years old
* American Society of Anesthesiologists (ASA) II-III
* Scheduled for posterolateral thoracotomy operation under general anesthesia

Exclusion Criteria:

* Patients with bleeding disorders,
* Mental or cognitive dysfunction
* History of chronic analgesic or drug abuse
* Allergy to local anesthetics
* Local infection at site of block

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
The degree of Postoperative Pain | 24 hours postoperative
  Postoperative pain will be assessed by the Numerical Rating Scale (NRS;0 no pain while 10 is the maximum pain) at 0,4,8,12,18, 24 hours during rest and cough. If the (NRS) is 4 or more, morphine 3mg will be titrated until pain relief is achieved using a short interval between boluses

SECONDARY OUTCOMES:
The amount of Postoperative morphine consumption | 24 hours Postoperative
  Total morphine consumption at 24 hours after surgery
Time to the first rescue analgesia request | 24 hours Postoperative
  Time till administration of first rescue analgesia
SpO2/FiO2 ratio | 24 hours Postoperative
  SpO2/FiO2 ratio at 6,8,12 and 24h postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Tanta University, Tanta, Elgarbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: For one year after completion of the study